CLINICAL TRIAL: NCT02596971
Title: A Phase IB/II Study Evaluating the Safety and Efficacy of Atezolizumab in Combination With Either Obinutuzumab Plus Bendamustine or Obinutuzumab Plus CHOP in Patients With Follicular Lymphoma or Rituximab Plus CHOP in Patients With Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Atezolizumab in Combination With Either Obinutuzumab Plus Bendamustine or Obinutuzumab Plus (+) Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP) in Participants With Follicular Lymphoma (FL) or Rituximab + CHOP in Participants With Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO29563; 2015-001364-19 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Diffuse Large B-Cell Lymphoma, Lymphoma Follicular
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — atezolizumab; Bendamustine Hydrochloride; Cyclophosphamide; Doxorubicin; obinutuzumab; Prednisone; Vincristine; Rituximab

ARMS (3):
- Atezo-G-Benda (Safety Run-In and Expansion Phases) (Experimental): Safety run-in phase: Participants with previously untreated or relapsed or refractory FL will receive obinutuzumab (G) and bendamustine during Cycle 1 (28-day cycle) and atezolizumab, obinutuzumab, and bendamustine during Cycles 2-6, during induction treatment, followed by atezolizumab (once monthly) and obinutuzumab (every other month [q2m]) for 24 months, during maintenance treatment. Expansion phase: Participants with previously untreated FL will receive same treatment regimen as described for safety run-in phase.
  Interventions: Drug: Atezolizumab; Drug: Bendamustine; Drug: Obinutuzumab
- Atezo-G-CHOP (Safety Run-In Phase) (Experimental): Safety run-in phase: Participants with previously untreated or relapsed or refractory FL will receive obinutuzumab and CHOP during Cycle 1 (21-day cycle) and atezolizumab, obinutuzumab, and CHOP during Cycles 2-6, during induction treatment, followed by atezolizumab (once monthly) and obinutuzumab (q2m) for 24 months, during maintenance treatment.
  Interventions: Drug: Atezolizumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Obinutuzumab; Drug: Prednisone; Drug: Vincristine
- Atezo-R-CHOP (Expansion Phase) (Experimental): Participants with previously untreated DLBCL will receive rituximab and CHOP during Cycle 1 (21-day cycle) and atezolizumab, rituximab, and CHOP during Cycles 2-8 (atezolizumab and rituximab for 8 cycles and CHOP for either 6 or 8 cycles, as determined by the investigator), during induction treatment, followed by atezolizumab from Cycles 9-25 during consolidation treatment.
  Interventions: Drug: Atezolizumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Vincristine; Drug: Rituximab

INTERVENTIONS:
Drug: Atezolizumab — Atezo-G-Benda: Atezolizumab 840 milligrams (mg) intravenously (IV) on Days 1 and 15 of Cycles 2-6, during induction treatment, followed by 840 mg IV on Days 1 and 2 of each month, starting with Month 1, during maintenance treatment. Atezo-G-CHOP: Atezolizumab 1200 mg IV on Day 1 Cycles 2-6, during induction treatment, followed by 840 mg IV on Days 1 and 2 of each month, starting with Month 1. Atezo-R-CHOP: Atezolizumab 1200 mg IV on Day 1 Cycles 2-8, during induction treatment, followed by 1200 mg IV on Day 1 of Cycles 9-25.
  Other Names: RO5541267; Tecentriq
Drug: Bendamustine — Bendamustine will be administered at a dose of 90 milligrams per square meter (mg/m^2) IV on Days 1 and 2 of Cycles 1-6, during induction treatment.
  Arms: Atezo-G-Benda (Safety Run-In and Expansion Phases)
Drug: Cyclophosphamide — Cyclophosphamide will be administered at a dose of 750 mg/m^2 IV on Day 1 of Cycle 1-6/8, during induction treatment.
  Arms: Atezo-G-CHOP (Safety Run-In Phase); Atezo-R-CHOP (Expansion Phase)
Drug: Doxorubicin — Doxorubicin will be administered at a dose of 50 mg/m^2 IV on Day 1 of Cycle 1-6/8, during induction treatment.
  Arms: Atezo-G-CHOP (Safety Run-In Phase); Atezo-R-CHOP (Expansion Phase)
Drug: Obinutuzumab — Atezo-G-Benda: Obinutuzumab will be administered at a dose of 1000 mg IV on Days 1, 8, and 15 of Cycle 1 and 1000 mg IV on Day 1 of Cycles 2-6, during induction treatment, followed by 1000 mg IV on Day 1 of every other month, starting with Month 1, during maintenance treatment. Atezo-G-CHOP: Obinutuzumab will be administered at a dose of 1000 mg IV on Days 1, 8, and 15 of Cycle 1 and 1000 mg IV on Day 1 of Cycles 2-6 during induction treatment, followed by 1000 mg IV on Day 1 of every other month, starting with Month 1 during maintenance treatment.
  Other Names: RO5072759
  Arms: Atezo-G-Benda (Safety Run-In and Expansion Phases); Atezo-G-CHOP (Safety Run-In Phase)
Drug: Prednisone — Prednisone will be administered at a dose of 40 mg/m^2 orally on Days 1-5 of Cycle 1-6/8, during induction treatment. Prednisolone may be given if prednisone is unavailable. The 40 mg/m^2 dose of prednisone on Day 1 will be replaced by oral corticosteroids given as premedication on Day 1 of Cycle 1 (and subsequent cycles).
  Arms: Atezo-G-CHOP (Safety Run-In Phase); Atezo-R-CHOP (Expansion Phase)
Drug: Vincristine — Vincristine will be administered at a dose of 1.4 mg/m^2 (maximum 2 mg) IV on Day 1 of Cycle 1-6/8, during induction treatment.
  Arms: Atezo-G-CHOP (Safety Run-In Phase); Atezo-R-CHOP (Expansion Phase)
Drug: Rituximab — Atezo-R-CHOP: Participants with previously untreated DLBCL will receive rituximab at a dose of 375 mg/m^2 IV on Day 1 of Cycle 1-8, during induction treatment.
  Arms: Atezo-R-CHOP (Expansion Phase)

SUMMARY:
This Phase Ib/II, open-label, multicenter, non-randomized study will evaluate the safety, efficacy, and pharmacokinetics of induction treatment consisting of atezolizumab in combination with either obinutuzumab + bendamustine (Atezo-G-benda) or obinutuzumab + CHOP (Atezo-G-CHOP) in participants with FL and atezolizumab + rituximab + chemotherapy (Atezo-R-CHOP) in participants with DLBCL, followed by post-induction treatment consisting of either atezolizumab plus obinutuzumab (Atezo-G) in participants with FL who achieve a complete response (CR) or partial response (PR) at end of induction (EOI) or atezolizumab alone in participants with DLBCL who achieve a CR at EOI.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* For participants enrolled in the safety run-in phase: lymphoma classified as either relapsed or refractory FL after treatment with at least one prior chemoimmunotherapy regimen or previously untreated Grade 1, 2, or 3a FL that requires treatment
* For participants enrolled in the expansion phase: lymphoma classified as either previously untreated Grade 1, 2, or 3a FL that requires treatment or previously untreated advanced DLBCL
* Histologically documented cluster of differentiation 20 (CD20) positive lymphoma
* Fluorodeoxyglucose-avid lymphoma
* At least one bi-dimensionally measurable lesion (greater than [>] 1.5 centimeters in its largest dimension by CT scan or magnetic resonance imaging)
* Availability of a representative tumor specimen and the corresponding pathology report for retrospective central confirmation of the diagnosis of FL or DLBCL
* For women who are not postmenopausal or surgically sterile: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than [<] 1 percent [%] per year during the treatment period and for at least 18 months after the last dose of study treatment for participants in the Atezo-G-benda and Atezo-G-CHOP treatment groups or for at least 12 months after the last dose of study treatment for participants in the Atezo-R-CHOP treatment group
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm

Exclusion Criteria:

* Histological evidence of transformation of FL into high-grade B-cell non-Hodgkin's lymphoma (NHL)
* Central nervous system lymphoma or leptomeningeal infiltration
* For participants with DLBCL: preplanned consolidative radiotherapy
* Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1
* For participants with relapsed or refractory FL: prior allogeneic or autologous stem cell transplantation, anthracycline therapy, treatment with fludarabine or alemtuzumab within 12 months prior to Day 1 of Cycle 1, treatment with a monoclonal antibody, radioimmunoconjugate, or antibody-drug conjugate within 4 weeks prior to Day 1 of Cycle 1, radiotherapy, chemotherapy, hormonal therapy, or targeted small-molecule therapy within 2 weeks prior to Day 1 of Cycle 1
* History of solid organ transplantation
* History of severe allergic or anaphylactic reaction or known sensitivity to humanized or murine monoclonal antibodies
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab, obinutuzumab, rituximab, or bendamustine formulation, including mannitol
* Positive for hepatitis B surface antigen (HBsAg), total hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) antibody at screening
* History of progressive multifocal leukoencephalopathy
* Vaccination with a live virus vaccine within 28 days prior to Day 1 of Cycle 1
* History of other malignancy, autoimmune disease, or any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results
* Major surgical procedure other than for diagnosis within 28 days prior to Day 1 of Cycle 1, or anticipation of a major surgical procedure during the course of the study
* For participants who will be receiving CHOP: left ventricular ejection fraction (LVEF) <50% by multiple-gated acquisition (MUGA) scan or echocardiogram
* Inadequate hematologic, renal, and liver function (unless due to underlying lymphoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- United States (9):
  - Rocky Mountain Cancer Center - Aurora, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University Miami, Miami, Florida
  - New York Uni Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oncology Associates of Oregon, P.C.; Willamette Valley Cancer Institute, Springfield, Oregon
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Texas Oncology, Austin, Texas
  - Texas Oncology-Tyler, Irving, Texas
- Australia (5):
  - Concord Repatriation General Hospital; Haematology, Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - The Queen Elizabeth Hospital; Haematology/Oncology, Woodville South, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
- Italy (7):
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna, Emilia-Romagna
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Emilia-Romagna
  - Az. Osp. S. Maria Delle Croci; U.O. Di Ematologia, Ravenna, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - AOU Città della Salute e della Scienza di Torino - Presidio Le Molinette, Torino, Lazio
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Azienda Ospedaliera Univ, Florence, Tuscany

REFERENCES:
- [Derived] Younes A, Burke JM, Cheson BD, Diefenbach CS, Ferrari S, Hahn UH, Hawkes EA, Khan C, Lossos IS, Musuraca G, Tani M, Vitolo U, Yuen S, Raval A, Shivhare M, Nielsen TG, Sellam G, Sharman JP. Safety and efficacy of atezolizumab with rituximab and CHOP in previously untreated diffuse large B-cell lymphoma. Blood Adv. 2023 Apr 25;7(8):1488-1495. doi: 10.1182/bloodadvances.2022008344. PMID 36287231
- [Derived] Younes A, Burke JM, Diefenbach C, Ferrari S, Khan C, Sharman JP, Tani M, Ujjani C, Vitolo U, Yuen S, Raval A, Shivhare M, Nielsen TG, Sellam G, Gilbertson M. Safety and efficacy of atezolizumab with obinutuzumab and bendamustine in previously untreated follicular lymphoma. Blood Adv. 2022 Oct 25;6(20):5659-5667. doi: 10.1182/bloodadvances.2021006131. PMID 35359000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 sites in 3 countries (Italy, Australia, and USA).
Pre-assignment Details: Out of the 117 subjects who were screened for this study, 91 subjects were enrolled to either FL treatment cohort (Atezo-G-Benda, Atezo-G-CHOP) or DLBCL cohort (Atezo-R-CHOP) and 26 subjects failed screening.
Groups:
- Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases): Safety run-in phase: Participants with previously untreated or relapsed or refractory FL received obinutuzumab (G) and bendamustine during Cycle 1 (28-day cycle) and atezolizumab, obinutuzumab, and bendamustine during Cycles 2-6, during induction treatment, followed by atezolizumab (once monthly) and obinutuzumab (every other month [q2m]) for 24 months, during maintenance treatment. Expansion phase: Participants with previously untreated FL received same treatment regimen as described for safety run-in phase.
- Atezo-G-CHOP Cohort (Safety Run-In Phase): Safety run-in phase: Participants with previously untreated or relapsed or refractory FL received obinutuzumab and CHOP during Cycle 1 (21-day cycle) and atezolizumab, obinutuzumab, and CHOP during Cycles 2-6, during induction treatment, followed by atezolizumab (once monthly) and obinutuzumab (q2m) for 24 months, during maintenance treatment.
- Atezo-R-CHOP Cohort (Expansion Phase): Participants with previously untreated DLBCL received rituximab and CHOP during Cycle 1 (21-day cycle) and atezolizumab, rituximab, and CHOP during Cycles 2-8 (atezolizumab and rituximab for 8 cycles and CHOP for either 6 or 8 cycles, as determined by the investigator), during induction treatment, followed by atezolizumab from Cycles 9-25 during consolidation treatment.
Period: Overall Study
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-G-CHOP Cohort (Safety Run-In Phase) | Atezo-R-CHOP Cohort (Expansion Phase)
Started | 42 | 7 | 42
Completed | 32 | 5 | 33
Not Completed | 10 | 2 | 9
Not completed — Death | 5 | 1 | 5
Not completed — Withdrawal by Subject | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Population: 3 populations for the Atezo-G-Benda cohort: safety, efficacy, and pharmacokinetic (PK). All participants (n = 42) in Atezo-G-Benda cohort included in safety and positron emission tomography (PET) evaluable populations. Two participants were excluded from efficacy evaluable population due to diagnosis of relapsed/ refractory follicular lymphoma (r/r FL). All 42 FL participants in Atezo-G-Benda cohort included in PK evaluable population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-G-CHOP Cohort (Safety Run-In Phase) | Atezo-R-CHOP Cohort (Expansion Phase) | Total
Number analyzed (Participants) | 42 | 7 | 42 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 6 | 20 | 61
  >=65 years | 7 | 1 | 22 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.9) | 57.4 (5.4) | 59.2 (15.7) | 57.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 4 | 16 | 40
  Male | 22 | 3 | 26 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 36 | 7 | 37 | 80
  Unknown or Not Reported | 3 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 37 | 6 | 40 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) at End of Induction (EOI), as Determined by the Independent Review Committee (IRC) Using Modified Lugano 2014 Criteria
Description: Primary end point was positron emission tomography (PET) CR at EOI by IRC according to modified Lugano classification using PET/CT scan. CR was defined as a score of 1 (no uptake above background), 2 (uptake less than or equal to [</=] mediastinum), or 3 (uptake less than [<] mediastinum but </=liver) with or without a residual mass on PET 5-point scale (5-PS), for lymph nodes and extralymphatic sites; no new lesions; no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow; and normal/immunohistochemistry (IHC)-negative bone marrow morphology. All PET evaluable 1L FL and 1L DLBCL participants with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Up to approximately 6 months
Population: Only Atezo-G-Benda and Atezo-R-Chop cohorts were evaluated for efficacy. 2 participants excluded from Atezo-G-Benda cohort (diagnosis of relapsed/refractory [r/r] FL). 2 participants excluded in R-Chop-Atezo cohort (they were excluded prior to Cycle 2, were not treated with atezolizumab).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 75 [61.29 to 85.76] | 77.5 [64.02 to 87.73]

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to approximately 4 years
Population: The safety analysis population consisted of all participants who received at least one dose of study drug. Safety analyses were based on the treatment that participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-G-CHOP Cohort (Safety Run-In Phase) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 42 | 7 | 42
percentage of participants | 100 | 100 | 100

3. Secondary Outcome: Percentage of Participants With CR at EOI, as Determined by the Investigator Using Lugano 2014 Criteria
Description: Tumor response assessment was performed by the investigator according to modified Lugano classification using PET/CT scan. CR was defined as a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. 90% confidence interval (CI) for percentage of responders was calculated using Clopper-Pearson method. All PET evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Up to approximately 6 months
Population: Only Atezo-G-Benda and Atezo-R-Chop cohorts were evaluated for efficacy. 2 participants excluded from Atezo-G-Benda cohort (diagnosis of r/r FL). 2 participants excluded in R-Chop-Atezo cohort (they were excluded prior to Cycle 2, were not treated with atezolizumab).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 87.5 [75.50 to 94.94] | 77.5 [64.02 to 87.73]

4. Secondary Outcome: Percentage of Participants With CR at EOI, as Determined by the IRC Using Modified Cheson 2007 Criteria
Description: Complete response according to the modified Cheson 2007 criteria using PET/CT scan: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy. Partial Response (PR): at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites; no increase in the size of the other nodes, liver, or spleen; with the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present. All PET evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 75.0 [61.29 to 85.76] | 77.5 [64.02 to 87.73]

5. Secondary Outcome: Percentage of Participants With CR at EOI, as Determined by the Investigator Using Modified Cheson 2007 Criteria
Description: Complete response according to modified Cheson 2007 criteria using PET/CT scan: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If bone marrow was involved by lymphoma prior to treatment, infiltrate must have cleared on repeat bone marrow biopsy. PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites; no increase in the size of other nodes, liver, or spleen; with exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present. All PET evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population. Only Atezo-G-Benda and Atezo-R-Chop cohorts were evaluated for efficacy.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 80.0 [66.80 to 89.64] | 75.0 [61.29 to 85.76]

6. Secondary Outcome: Percentage of Participants With Objective Response (CR or PR) at EOI, as Determined by the IRC Using Modified Cheson 2007 Criteria
Description: Objective response: having CR or PR as assessed according to the modified response criteria for iNHL (Modified Cheson et al, 2007). CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy. PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites; no increase in the size of the other nodes, liver, or spleen; with the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present. All positron emission tomography (PET) evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 90.0 [78.56 to 96.51] | 90.0 [78.56 to 96.51]

7. Secondary Outcome: Percentage of Participants With Objective Response (CR or PR) at EOI, as Determined by the Investigator Using Modified Cheson 2007 Criteria
Description: as for outcome 6
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 95.0 [85.08 to 99.10] | 87.5 [75.50 to 94.94]

8. Secondary Outcome: Percentage of Participants With Objective Response (CR or PR) at EOI, as Determined by the IRC Using Lugano 2014 Criteria
Description: Tumor response assessment was performed by IRC according to modified Lugano classification using PET/CT scan. OR defined as a response of CR or PR. CR: a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with/without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. PR: a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites; no new lesions; and reduced residual uptake in bone marrow compared with baseline. All positron emission tomography (PET) evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 90.0 [78.56 to 96.51] | 87.5 [75.50 to 94.94]

9. Secondary Outcome: Percentage of Participants With Objective Response (CR or PR) at EOI, as Determined by the Investigator Using Lugano 2014 Criteria
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using PET/CT scan. OR: a response of CR or PR. CR: a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes & extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. PR with a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites; no new lesions; and reduced residual uptake in bone marrow compared with baseline. All positron emission tomography (PET) evaluable 1L FL and 1L DLBCL patients with at least one dose of atezolizumab were included in efficacy population.
Time Frame: Up to approximately 6 months
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 95.0 [85.08 to 99.10] | 87.5 [75.50 to 94.94]

10. Secondary Outcome: Percentage of Participants With Best Response of CR or PR During Study, as Determined by Investigator Using Modified Cheson 2007 Criteria
Description: CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy, liver and spleen have returned to normal size (if enlarged at baseline), If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy. PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites; no increase in the size of the other nodes, liver, or spleen; with the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present. Only Atezo-G-Benda and Atezo-R-Chop cohorts were evaluated for efficacy.
Time Frame: Baseline up to approximately 4 years (assessed at Baseline, 6 to 8 weeks after Day [D] 1 of Cycle [Cy] 6 or 8 (1Cy: 21 or 28 days), then every 2 months up to 24 months, at 35 days of last dose, and at every 3 months post-treatment follow-up [up 4 years])
Population: All PET evaluable 1L FL and 1L DLBCL patients that received at least one dose of atezolizumab.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 40 | 40
percentage of participants | 80.0 [66.80 to 89.64] | 75.0 [61.29 to 85.76]

11. Secondary Outcome: Observed Serum Obinutuzumab Concentration
Description: Predose time point was "any time prior to dose" for Cycle (Cy) 1 and "within 5 hour prior to dose" for other cycles (Cy 2,5,6) and for Months 1 to 24 during maintenance phase. Infusion duration for administration of first infusion should begin at an initial rate of 50 milligrams per hour (mg/hour). If no reaction occurs, increase the infusion rate in 100 mg/hour increments every 30 minutes to a maximum of 400 mg/hour.
Time Frame: Induction: Predose, 0.5 hour (h) postinfusion on Day (D) 1 of Cy1,2,5,6 (1Cy: 21/28 days); Maintenance: Predose, 0.5h postinfusion on Day 1 of Month 1,3,7,15,23; 120 days & 1 year of last dose or at treatment discontinuation (up to 4 years)
Population: All participants who received at least 1 dose of study treatment and who provided at least one pharmacokinetic (PK) sample.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-G-CHOP Cohort (Safety Run-In Phase)
Number analyzed (Participants) | 42 | 7
ug/mL
  C1 Cmax after 1st infusion: number analyzed (Participants) | 35 | 5
  C1 Cmax after 1st infusion | 329 [21.7 to 513] | 400 [284 to 450]
  C1 Cmin after the last infusion on C1: number analyzed (Participants) | 39 | 7
  C1 Cmin after the last infusion on C1 | 322 [168 to 486] | 399 [236 to 611]
  C6 - Cmax after last dosing of induction: number analyzed (Participants) | 20 | 7
  C6 - Cmax after last dosing of induction | 544 [387 to 883] | 659 [287 to 838]
  C6 - Cmin after last dosing of induction: number analyzed (Participants) | 22 | 7
  C6 - Cmin after last dosing of induction | 203 [137 to 471] | 245 [171 to 481]

12. Secondary Outcome: Observed Serum Atezolizumab Concentration
Description: Atezo-G-Benda: Induction:Predose on D1 of Cy5,6 & D1,15 of Cy2,3 (1Cy:21/28 days), Cy2D1:0.5h postinfusion; Maintenance:Predose on D1 of Month 1,2,4,7,15,23, Month 2 D1: 0.5h postinfusion; 120 days & 1 year of last dose or at treatment discontinuation (up to 4 years); Atezo-G-CHOP: Induction:Predose on D1 of Cy2,3,5,6 (1Cy:21 days), Cy2D1:0.5h postinfusion; Maintenance:Predose on D1 of Month 1,2,3,4,7,15,23, Month 2 D1: 0.5h postinfusion; 120 days & 1 year of last dose or at treatment discontinuation (up to 4 years). Predose time point was "within 5 hour prior to dose" for Cy2,3,5,6 during induction phase and for Months 1 to 24 during maintenance phase. infusion length: 30-60 minutes.
Time Frame: Atezo-R-CHOP: Predose on D1 of Cy2,3,5,8,9,10,11,12,16,20,25 (1Cy:21 days), 0.5h postinfusion of D1 of Cy2,9; at 120 days & 1 year of last dose or at treatment discontinuation (up to 4 years)
Population: All participants who received at least 1 dose of study treatment and who provided at least one pharmacokinetic (PK) sample. 0 represents no data was collected at that cycle.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-R-CHOP Cohort (Expansion Phase) | Atezo-G-CHOP Cohort (Safety Run-In Phase)
Number analyzed (Participants) | 42 | 42 | 7
ug/mL
  Cycle 2 - Cmax after 1st infusion: number analyzed (Participants) | 31 | 31 | 7
  Cycle 2 - Cmax after 1st infusion | 275 [193 to 388] | 332 [227 to 472] | 424 [340 to 670]
  C2 - Cmin before 2nd infusion: number analyzed (Participants) | 32 | 34 | 6
  C2 - Cmin before 2nd infusion | 83 [59 to 128] | 82.1 [55.7 to 122] | 94 [65 to 139]
  C6 - Cmin after 6th infusion: number analyzed (Participants) | 20 | 0 | 6
  C6 - Cmin after 6th infusion | 256 [93 to 369] |  | 195 [157 to 296]
  C8 - Cmax after 7th infusion: number analyzed (Participants) | 0 | 22 | 0
  C8 - Cmax after 7th infusion |  | 486.5 [363 to 793] |
  C8 - Cmin before 8th infusion: number analyzed (Participants) | 0 | 23 | 0
  C8 - Cmin before 8th infusion |  | 184 [104 to 359] |

13. Secondary Outcome: Observed Serum Rituximab Concentration
Description: Predose time point was "any time prior to dose" for Cycle 1 and "within 5 hour prior to dose" for other cycles (Cycles 2,5,8) during induction phase and for Months 1 to 24 during maintenance phase. Infusion duration for administration of first infusion should begin at an initial rate of 50 mg/hour. If no infusion-related or hypersensitivity reaction occurs, increase the infusion rate in 50 mg/hour increments every 30 minutes to a maximum of 400 mg/hour. If no reaction occurs, increase the infusion rate in 100 mg/hour increments every 30 minutes to a maximum of 400 mg/hour.
Time Frame: Predose, 0.5h postinfusion on D1 of Cy1,2,5,8 (1Cy: 21 days); at 120 days and 1 year after last rituximab dose or at treatment discontinuation (up to 4 years)
Population: All participants who received at least 1 dose of study treatment and who provided at least one PK sample.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 42
ug/mL
  C1 - Cmax after dosing C1: number analyzed (Participants) | 34
  C1 - Cmax after dosing C1 | 159 [0.5 to 292]
  C1 - Ctrough after dosing C1: number analyzed (Participants) | 34
  C1 - Ctrough after dosing C1 | 26.1 [0.5 to 41.3]
  C8 - Cmax after dosing C8: number analyzed (Participants) | 27
  C8 - Cmax after dosing C8 | 229 [185 to 303]
  C8 - Ctrough after dosing C8: number analyzed (Participants) | 26
  C8 - Ctrough after dosing C8 | 105.5 [39.9 to 150]

14. Secondary Outcome: Percentage of Participants With Human Anti-Human Antibodies (HAHAs) to Obinutuzumab
Description: Induction: Predose (any time prior to dose) on D1 of Cy1,5,6 (1Cy: 21/28 days); Maintenance: Predose (any time prior to dose) on D1 of Month 1; at 120 days and 1 year of last obinutuzumab dose or at treatment discontinuation (up to 4 years)
Time Frame: Baseline up to approximately 4 years
Population: The safety analysis population consisted of all participants who received at least one dose of study drug in the Atezo-G-Benda cohort
Measure: Number; unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases)
Number analyzed (Participants) | 42
percentage of participants
  Induction Cycle 1 Day 1 | 2.4
  Induction Cycle 5 Day 1: number analyzed (Participants) | 31
  Induction Cycle 5 Day 1 | 0
  Induction Cycle 6 Day 1: number analyzed (Participants) | 34
  Induction Cycle 6 Day 1 | 0
  Maintenance Month 1: number analyzed (Participants) | 37
  Maintenance Month 1 | 0
  Study Drug Completion or Early Discontinuation: number analyzed (Participants) | 14
  Study Drug Completion or Early Discontinuation | 0
  Obinutuzumab Day 120 Follow up: number analyzed (Participants) | 33
  Obinutuzumab Day 120 Follow up | 0

15. Secondary Outcome: Percentage of Participants With Human Anti-Chimeric Antibodies (HACAs) to Rituximab
Description: Induction: Predose (any time prior to dose) on D1 of Cy1,5,8 (1Cy: 21 days); Maintenance: at 120 days and 1 year of last rituximab dose or at treatment discontinuation (up to 4 years)
Time Frame: Baseline up to approximately 4 years
Population: The safety analysis population consisted of all participants who received at least one dose of study drug in the Atezo-R-CHOP cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 42
percentage of participants
  Baseline: number analyzed (Participants) | 35
  Baseline | 14.3
  Induction Cycle 1 Day 1: number analyzed (Participants) | 2
  Induction Cycle 1 Day 1 | 0
  Induction Cycle 5 Day 1: number analyzed (Participants) | 36
  Induction Cycle 5 Day 1 | 0
  Induction Cycle 8 Day 1: number analyzed (Participants) | 28
  Induction Cycle 8 Day 1 | 0
  Rituximab Day 120 Follow up: number analyzed (Participants) | 6
  Rituximab Day 120 Follow up | 0
  Rituximab 1 Year Follow up: number analyzed (Participants) | 11
  Rituximab 1 Year Follow up | 0
  Study Drug Completion or Early Discontinuation: number analyzed (Participants) | 13
  Study Drug Completion or Early Discontinuation | 0

16. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezolizumab
Description: Atezo-G-CHOP: Induction: Predose on D1 of Cy2,3,5,6 (1 Cy: 21 days); Maintenance: Predose on D1 of Month 1,2,4,7,15,23; at 120 days and 1 year of last atezolizumab dose or at treatment discontinuation (up to 4 years); Atezo-R-CHOP: Predose on D1 of Cy 2,3,5,8,16,25 (1 Cy: 21 days); at 120 days and 1 year of last atezolizumab dose or at treatment discontinuation (up to 4 years). Predose time point was "any time prior to dose" for Cycles 2,3,5,6,8 during induction phase, for Cycles 16,25 during consolidation treatment, and for Months 1 to 24 during maintenance phase. Atezo-G-Benda: Induction: Predose on D1 of Cy2,3,5,6 (1Cy: 28 days), Cy3D15: Predose; ; Maintenance: Predose on D1 of Month 1,4,7,15,23; at 120 days and 1 year of last atezolizumab dose or at treatment discontinuation (up to 4 years). The percentage of participants with positive results for ATAs to atezolizumab at baseline and at post-baseline time points are reported.
Time Frame: Baseline up to approximately 4 years
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-G-CHOP Cohort (Safety Run-In Phase) | Atezo-R-CHOP Cohort (Expansion Phase)
Number analyzed (Participants) | 42 | 7 | 42
percentage of participants
  Baseline: number analyzed (Participants) | 42 | 7 | 35
  Baseline | 2.4 | 0 | 14.3
  Induction Cycle 2 Day 1: number analyzed (Participants) | 41 | 7 | 39
  Induction Cycle 2 Day 1 | 0 | 0 | 2.6
  Consolidation Cycle 16: number analyzed (Participants) | 0 | 0 | 17
  Consolidation Cycle 16 |  |  | 5.9
  Atezolizumab Day 120 Follow up: number analyzed (Participants) | 17 | 2 | 11
  Atezolizumab Day 120 Follow up | 0 | 0 | 9.1
  Atezo PK and Immunogenicity Follow Up (1YR): number analyzed (Participants) | 12 | 4 | 18
  Atezo PK and Immunogenicity Follow Up (1YR) | 0 | 0 | 5.6

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 4 years
Description: The safety population is defined as all patients who received at least one dose of the study medication.
Arm/Group | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) | Atezo-G-CHOP Cohort (Safety Run-In Phase) | Atezo-R-CHOP Cohort (Expansion Phase)
All-Cause Mortality (participants affected / at risk) | 5/42 | 1/7 | 5/42
Serious Adverse Events (participants affected / at risk) | 19/42 | 2/7 | 18/42
Other Adverse Events (participants affected / at risk) | 42/42 | 7/7 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) (N=42) | Atezo-G-CHOP Cohort (Safety Run-In Phase) (N=7) | Atezo-R-CHOP Cohort (Expansion Phase) (N=42)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 6 (7)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
IMMUNE-MEDIATED ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 3 (3) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 0 (0) | 2 (2)
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PROGRESSIVE MULTIFOCAL LEUKOENCEPHALOPATHY (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OBLITERATIVE BRONCHIOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezo-G-Benda Cohort (Safety Run-In and Expansion Phases) (N=42) | Atezo-G-CHOP Cohort (Safety Run-In Phase) (N=7) | Atezo-R-CHOP Cohort (Expansion Phase) (N=42)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 6 (8)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 14 (22) | 3 (6) | 22 (31)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (6) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
HYPOPHYSITIS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 1 (1) | 2 (2)
DRY EYE (Eye disorders) | 2 (2) | 2 (2) | 3 (3)
OCULAR HYPERAEMIA (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 3 (3) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (10) | 2 (3) | 5 (5)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (7) | 0 (0) | 4 (4)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 18 (27) | 3 (4) | 18 (26)
DEFAECATION URGENCY (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 20 (47) | 3 (10) | 14 (23)
DRY MOUTH (Gastrointestinal disorders) | 5 (5) | 0 (0) | 4 (4)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 8 (11) | 1 (1) | 2 (3)
FLATULENCE (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
GLOSSITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 22 (42) | 5 (8) | 13 (22)
RECTAL DISCHARGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
STEATORRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (5)
VOMITING (Gastrointestinal disorders) | 11 (15) | 2 (3) | 9 (11)
ASTHENIA (General disorders) | 3 (5) | 0 (0) | 2 (4)
CHEST DISCOMFORT (General disorders) | 2 (2) | 1 (1) | 2 (2)
CHEST PAIN (General disorders) | 10 (10) | 1 (1) | 4 (4)
CHILLS (General disorders) | 3 (5) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 23 (27) | 5 (6) | 17 (22)
FEELING COLD (General disorders) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 7 (9) | 1 (1) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 1 (2) | 2 (3) | 3 (5)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 1 (1) | 3 (4)
PAIN (General disorders) | 2 (2) | 1 (1) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 3 (3) | 1 (2) | 1 (1)
PYREXIA (General disorders) | 10 (12) | 0 (0) | 5 (9)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 3 (5) | 0 (0) | 2 (2)
BRONCHITIS (Infections and infestations) | 4 (4) | 1 (2) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 5 (8) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
SINUSITIS (Infections and infestations) | 7 (7) | 1 (1) | 5 (5)
SKIN INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 (22) | 1 (1) | 7 (7)
URINARY TRACT INFECTION (Infections and infestations) | 6 (8) | 1 (1) | 1 (2)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (5)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 29 (45) | 2 (2) | 16 (16)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
AMYLASE INCREASED (Investigations) | 4 (4) | 0 (0) | 3 (3)
LIPASE INCREASED (Investigations) | 13 (14) | 1 (1) | 4 (6)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (4) | 9 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (6) | 8 (13)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1) | 4 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0) | 2 (2)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (2) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 4 (4)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 5 (5)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (10) | 1 (1) | 2 (2)
ACROCHORDON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
AMNESIA (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 7 (12) | 1 (1) | 4 (6)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6)
HEADACHE (Nervous system disorders) | 19 (25) | 1 (1) | 8 (13)
HYPOAESTHESIA (Nervous system disorders) | 4 (4) | 2 (3) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 3 (5) | 0 (0) | 3 (3)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 (3) | 2 (3) | 13 (15)
TASTE DISORDER (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3)
DEVICE OCCLUSION (Product Issues) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 7 (7) | 0 (0) | 3 (6)
INSOMNIA (Psychiatric disorders) | 7 (7) | 2 (2) | 7 (8)
MANIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (3) | 1 (1) | 1 (1)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
VULVOVAGINAL PAIN (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 25 (31) | 5 (9) | 12 (18)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1) | 3 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 1 (1) | 4 (4)
PHARYNGEAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 5 (6)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 10 (10)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 12 (14) | 0 (0) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 14 (22) | 0 (0) | 4 (6)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0)
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 6 (9) | 0 (0) | 1 (1)
PERIPHERAL COLDNESS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Development of the atezolizumab combination treatment was discontinued as there was insufficient evidence regarding the additive efficacy of this therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT02596971/Prot_SAP_001.pdf